CLINICAL TRIAL: NCT01374061
Title: Pre Hospital Evaluation of Video Laryngoscopy : a Comparative Study of Macintosh and GLIDESCOPE Ranger®
Brief Title: Pre Hospital Evaluation of Video Laryngoscopy
Acronym: EVE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100205; 2010-A01512-37 (Other: IDRCB)
Record Dates: First submitted 2011-05-25; First posted 2011-06-15 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Cardiac Arrest; Respiratory Distress Syndrome; Shock; Acute Post-trauma Stress State; Drug Toxicity; Trauma, Nervous System
Keywords: Emergency intubation; Glide scope Ranger; Pre hospital
MeSH Terms: conditions — Heart Arrest; Respiratory Distress Syndrome; Shock; Drug-Related Side Effects and Adverse Reactions; Trauma, Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Classical intubation (Active Comparator)
  Interventions: Device: Classical intubation
- 2: Glidescope intubation (Experimental)
  Interventions: Device: GLIDESCOPE

INTERVENTIONS:
Device: Classical intubation — Classical intubation
  Arms: 1: Classical intubation
Device: GLIDESCOPE — GLIDESCOPE intubation
  Arms: 2: Glidescope intubation

SUMMARY:
The objective of this work is to compare standard intubation with video laryngoscope (Glide scope Ranger ) in French pre hospital multicentric study.

DETAILED DESCRIPTION:
Introduction: In France, patients in critical status brought to hospital by emergency physicians and nurses experimented in tracheal intubation. It is an invasive act allowing a protection of airways and an optimal oxygenation of the patients in distress. The reference technique is the direct laryngoscopy by Macintosh . Corresponding data shows that a video laryngoscope - GLIDESCOPE laryngoscope - improve the conditions of intubation in the surgical unit thanks to a better display(visualization) of the opening. A derived device for pre hospital emergency units (GLIDESCOPE Ranger®) deserves to be compared with the classic laryngoscopy in emergency conditions.

Objectives: compare the emergency intubation in Pre hospital meadow by Glide Scope Ranger with regard to the classic method

Progress of the study: the patients will be included by emergency physicians working in out of hospital teams of 3 major hospitals of Paris. The patients will be randomized in 2 groups: 1 group classic laryngoscopy (group 1) and a group Glide scope Ranger (group 2). The score IDS will be compared for every group as well as the arisen of a complication during the procedure. The consent will be collected on the place or during the hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* patients of more than 18 years old
* requiring an intubation
* by medical out of hospital emergency operators
* medical insurance
* Consent signed

Exclusion Criteria:

* Age <18, pregnant women
* Refusal of consent or inability for understanding study
* small mouth opening makes it impossible intubate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
IDS score in each group | during the intubation

SECONDARY OUTCOMES:
Vomit / regurgitation or inhalation per-procedure | during the intubation
Dental or throat traumatism | during the intubation
Broncho/laryngospasm | during the intubation
Hypoxia | per intubation
Hemodynamic instability | per intubation
Inhalation pneumonia | within 24 hours following the inclusion
Failure of intubate | during the intubation

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GALLULA, Ph, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Patrick PLAISANCE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris